CLINICAL TRIAL: NCT05103995
Title: Impact of Donor-recipient ABO Matching on Patients' Outcome After Peripheral Blood Stem Cell Haploidentical Stem Cell Transplantation
Brief Title: Impact of Donor-recipient ABO Matching on Haploidentical Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Affiliated Jinhua Hospital of Zhejiang University (Unknown)
Responsible Party: Principal Investigator, Yi Luo, Principal Investigator, First Affiliated Hospital of Zhejiang University
Other Study IDs: ZJU-haplo-abo
Record Dates: First submitted 2021-10-10; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Hematological Malignancies; Haploidentical Stem Cell Transplantation
Keywords: haploidentical stem cell transplantation; hematological malignancies; ABO incompatibility
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ABO matched: Donor-recipient ABO matched
  Interventions: Other: no intervention
- Minor incompatibility: Donor-recipient minor incompatibility
  Interventions: Other: no intervention
- Major incompatibility: Donor-recipient major incompatibility
  Interventions: Other: no intervention
- Bidirectional incompatibility: Donor-recipient bidirectional incompatibility
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, just observation

SUMMARY:
the impact of donor-recipient ABO matching on outcome of peripheral blood stem cell haploidentical hematopoietic stem cell transplantation

DETAILED DESCRIPTION:
The impact of donor-recipient ABO compatibility on transplant outcomes had been evaluated in different transplant settings, but had shown different results. The investigators set out to investigate the impact of ABO incompatibility on post-transplant outcomes, engraftment kinetics and blood product requirements, transfusion independence, the incidence of poor graft function (PGF) in anti-T-lymphocyte globulin (ATG) based haplo-SCT with PBSC grafts.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects or their legal representatives signed the informed consent before the clinical study. 2. Subjects aged 15-70 years. 3. Patients with malignant hematological diseases plan to receive allogeneic peripheral blood stem cell transplantation 4. Patients have no suitable HLA identical sibling donor 5.Patients with malignant hematological diseases plan to receive HLA haploidentical stem cell transplantation 6. Subjects with ECoG score of 0-2.

Exclusion Criteria:

1.Patients have suitable HLA identical sibling donor 2. Patients with severe liver and kidney function (alanine aminotransferase > 2.5 times of the upper normal limit, serum creatinine > 1.5 times of the upper normal limit), cardiopulmonary dysfunction (cardiac function NYHA III / IV, cardiac ejection fraction < 50%, severe obstructive or restrictive ventilation dysfunction); 3. Patients with active infection; 4. patients diagnosed with aplastic anemia before transplantation or died within 2 months after transplantation; 5. Subjects with ECoG score > 2; 6. Patients with secondary tumor; 7. Patients who cannot independently choose to enter or exit clinical trials due to serious central nervous system disease or mental disease.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with malignant hematological diseases plan to receive allogeneic peripheral blood stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
5-year Overall Survival | 5 year
  5-year Overall Survival

SECONDARY OUTCOMES:
5-year Non-relapse mortality | 5 year
  5-year non-relapse mortality
5-year cumulative incidence of chronic graft versus host disease | 5 year
  5-year cumulative incidence of chronic graft versus host disease
28-day cumulative incidence of neutrophils engraftment | 28 day
  numbers of participants achieved neutrophils engraftment at 28 days post transplantation
28-day cumulative incidence of platelets engraftment | 28 day
  numbers of participants achieved platelets engraftment at 28 days post transplantation
365-day blood transfusion requirements | 365 day
  numbers of blood products transfusion within 365-day after transplantation
cumulative incidence of blood transfusion independence within 60 days after transplantation | 60 day
  numbers of participants achieved blood transfusion independence within 60 days after transplantation
the 5-year cumulative incidence of poor graft function the incidence of poor graft function | 5 year
  numbers of participants occurred poor graft function 5 years post transplantation
the 5-year cumulative incidence of graft failure | 5-year
  numbers of participants occurred graft failure 5 years post transplantation
100-day cumulative incidence of acute graft versus host disease | 100-day
  100-day cumulative incidence of acute graft versus host disease

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The first Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Affiliated Jinhua hospital of Zhejiang University, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No